CLINICAL TRIAL: NCT04846465
Title: Femoral Neck-shaft Angle in Sohag Population: Variation Relating to Age and Sex.
Brief Title: Femoral Neck-shaft Angle in Sohag Population
Acronym: NSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marina Talaat Bushra, Demonstrator at Anatomy and Embryology Department Faculty of Medicine -Sohag University, Sohag University
Other Study IDs: Soh-Med-21-04-05
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Hip Abnormalities; Femur; Angulation; Urinary Stone; Lower Limb Arterial Embolus
MeSH Terms: conditions — Urinary Calculi | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- male: normal Sohag healthy male (≥18 & ≤ 60 years)
  Interventions: Other: Screening in picture archiving and communication system (PACS) .
- female: normal Sohag healthy female (≥18 & ≤ 60 years)
  Interventions: Other: Screening in picture archiving and communication system (PACS) .

INTERVENTIONS:
Other: Screening in picture archiving and communication system (PACS) . — Screening in picture archiving and communication system (PACS) , the images of the participants who underwent computed tomography (CT) of the femur and acetabulum.

SUMMARY:
The femur or thigh bone is the strongest and longest bone of the body and about 45 cm long in an average man that means approximately one fourth of the height of individual. It has upper end, lower end and a cylindrical shaft. Upper end consists of head, neck. The neck is about 5 cm long, connects the head to the shaft and is directed upward, medially and slightly forward and making an angle about 125 with shaft but the angle is wider in children. The neck-shaft angle (NSA ) is defined as the angle formed by the neck axis and long axis of the shaft of femur.The knowledge of the neck shaft angle is valuable in the diagnosis and treatment of fracture of upper end of femur.

The aim of the study is :

1. to evaluate the normal values of femoral neck-shaft angle
2. to detect factors that may affect this angle as age, and sex, in Egyptian adults from Sohag.

ELIGIBILITY:
Inclusion Criteria:

* Adults, eligible and adequate imaging data for measurement, and absence of fracture, arthritis, tumor, deformity, or surgery on the proximal part of the femur or any disorder that may affect measurements of femoral neck-shaft angle

Exclusion Criteria:

* Adults with incomplete imaging data; and fracture, arthritis, tumor, deformity, or surgery on the proximal part of the femur

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants who underwent computed tomography (CT) of the femur and acetabulum in departments of Radiology in Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-14 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
To measure femoral neck-shaft angle ( NSA) . | 16 weeks following the startpoint of the study
  We will use Computed Tomography (CT) in determination and measurement of femoral neck shaft angle ( NSA) and its variation relating to age and sex.
  Neck-shaft angle will be measured using Image Works by noting angle between two intersection lines representing proximal femoral shaft axis and the femoral neck axis.
  Normal neck-shaft angle varies from 115°-140° (mean of 126°). Normal range neck shaft angle is 121°-138°in male. Normal range neck shaft angle is 119°-137°in female.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt